CLINICAL TRIAL: NCT04386889
Title: SLE Vasculitis Incidence In Female Egyptian Patients
Brief Title: SLE Vasculitis In Egyptian Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tabarak New Cairo Hospital (TNCH) (Other)
Responsible Party: Principal Investigator, Prof. Dr. /Tayseer Abdulaal, Prof. Dr., Tabarak New Cairo Hospital (TNCH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SLE Tabarak 01
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Vasculitis Lupus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SLE Vasculitis (Other): 20 SLE Female patients will subjected to study of the all vasculitic pattern that may occur.
  Interventions: Other: Vasculitis In SLE

INTERVENTIONS:
Other: Vasculitis In SLE — 20 SLE female Egyptian patients, among them we are going to study the vasculitic pattern incidence.

SUMMARY:
Systemic lupus erythematosus (SLE) is a complex heterogeneous autoimmune disease with a wide variety of clinical and serological manifestations that may affect any organ. Vasculitis prevalence in SLE is reported to be between 11% and 36%.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a complex heterogeneous autoimmune disease with a wide variety of clinical and serological manifestations that may affect any organ. Vasculitis prevalence in SLE is reported to be between 11% and 36%. A diverse clinical spectrum, due to inflammatory involvement of vessels of all sizes, is present. Even though cutaneous lesions, representing small vessel involvement, are the most frequent, medium and large vessel vasculitis may present with visceral affection, with life-threatening manifestations such as mesenteric vasculitis, pulmonary hemorrhage, or mononeuritis multiplex, with detrimental consequences. Early recognition and an appropriate treatment are crucial. Recent studies have shown that vasculitis in patients with SLE may present different clinical forms based on the organ involved and the size of the affected vessel. It is noteworthy that the episodes of vasculitis are not always accompanied by high disease activity. Recent articles on this topic have focused on new treatments for the control of vascular disease, such as biological therapies such as Rituximab and Belimumab, among others.

ELIGIBILITY:
Inclusion Criteria:

* LE or suspected SLE established by ACR criteria
* Ability to give informed consent
* Adult and minor relatives (first and second degree) of individuals Included in IV-G (only for genetic studies)
* Ability of the patient or minor relative s parents to give informed consent
* Affected individuals age greater than or equal to 9 years with no upper age limit
* Healthy Volunteers (non-related) age greater than or equal to 18 with no upper age limit
* Healthy Volunteers (first- and second-degree relatives) age greater than or equal to 9 with no upper age limit
* Vascular studies adults only age greater than or equal to 18 with no upper age limit

Exclusion Criteria:

* Concomitant medical problems which would confound the interpretation of studies gathered by this protocol. Included in this is the presence of HIV in the blood, active malignancies, or other significant medical conditions that may interferes with interpretation of some lupus studies.
* Concomitant medical, surgical or other conditions for which inadequate facilities are available to support their care at NIH.

Inability or unwillingness to comply with follow up requirements (e.g. distance, social, physical limitations)

* Any comorbidity of medical or psychological/psychiatric condition or treatment after reviewing of patients previous or outside medical records, that in the opinion of the Principal Investigator, would exclude the subjects from the research studies (e.g. Patient requiring urgent and/or acute medical care, surgical or other procedures)
* Unwilling to participate in research studies or to provide research samples or data.

Criteria for exclusion:

- Any concomitant medical problems or are taking medications which would confound the interpretation of studies they are considered for

EXCLUSION CRITERIA FOR VASCULAR STUDIES ONLY, FOR SLE AND HEALTHY CONTROLS:

* Subjects with a contraindication to MRI scanning will not receive the optional Cardiovascular MRI. These contraindications include subjects with the following devices:
* Central nervous system aneurysm clips unless it is labeled safe or conditional for MRI
* Implanted neural stimulator (e.g.TENS-Unit) unless it is labeled safe or conditional for MRI
* Implanted cardiac pacemaker or defibrillator
* Cochlearor any type of ear implant unless it is labeled safe or conditional for MRI
* Ocular foreign body (e.g. metal shavings)
* Implanted Insulin pump or drug infusion device unless it is labeled safe or conditional for MRI
* Metal shrapnel or bullet unless cleared by plain x-ray as safe for MRI
* Subjects with renal excretory dysfunction, estimated glomerular filtration rate < 60 mL/min/1.73m(2) using the CKD-EPI equation or equivalent (using the CRIS-calculated eGFR to define the threshold) and a serum creatinine measured within 2 weeks without intercurrent change in medical condition or medications. Subjects meeting this exclusion criterion may still be included in the study but will not be exposed to the cardiac CT angiography, or gadolinium-based contrast agents.
* Any clinical instability precluding subject from getting MRI as determined by the enrolling clinician.
* Pregnant or lactating women will be excluded from vascular studies.
* Healthy controls with known history of coronary artery disease, peripheral vascular disease or atherosclerosis.
* Individuals younger than 18 years old will be excluded given the radiation exposure as well as the lack of proper validation for the proposed vascular function studies.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-25 (Estimated); Primary Completion 2021-07-25 (Estimated); Study Completion 2021-08-25 (Estimated)

PRIMARY OUTCOMES:
SLE Vasculitis | 6 months
  Incidence of vasculitic pattern

CONTACTS AND LOCATIONS:
Locations (1):
- Tabarak New Cairo Hospital, Cairo, Egypt